CLINICAL TRIAL: NCT02215772
Title: A Phase I Trial to Investigate the Metabolism and Pharmacokinetics of an Open Label Single Dose of 200 mg [14C]-BI 44370 BS Administered as an Oral Solution in Healthy Male Volunteers
Brief Title: Metabolism and Pharmacokinetics of [14C]-BI 44370 BS Administered as an Oral Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1246.14
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (1):
- BI 44370 BS (Experimental): 200 mg containing 2.43 megabecquerel (MBq) 14C-radioactivity
  Interventions: Drug: BI 44370 BS

INTERVENTIONS:
Drug: BI 44370 BS

SUMMARY:
Study to investigate the basic pharmacokinetics of BI 44370 BS, its metabolite CD 10419 BS, and 14C-radioactivity including mass balance, excretion pathways, and metabolism following a single oral administration of 200 mg [14C]BI 44370 BS to healthy male volunteers and to evaluate safety and tolerability following a single oral administration of 200 mg [14C]BI 44370 BS to healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG, clinical laboratory tests
* Age ≥18 and ≤65 years
* Body mass index (BMI) ≥18.0 and BMI ≤30.0 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic, or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to study drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration until after the last sample from Visit 2 is collected
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking during the stay in the trial centre
* Alcohol abuse (more than on average 2 units of alcoholic beverages per day or more than 14 units per week (1 unit equals 1 pint [285 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit))
* Drug abuse
* Blood donation (more than 100 mL within 60 days prior to study drug administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial until follow-up examination)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* Veins unsuitable for blood sampling
* PR interval >220 ms or QRS interval >120 ms
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a medical trial in the previous year
* Irregular defecation pattern (less than once per 2 days)
* Not willing to use adequate contraception (condoms use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until three months after the last intake

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Individual time course profiles of [14C]-radioactivity in whole blood, plasma, urine | up to day 15
  in nmoleq/L
Individual time course profiles of [14C]-radioactivity in faeces | up to day 15
  in nmoleq/kg
Individual time course profiles of BI 44370 BS (and its glucuronide CD 10419 BS) in plasma and urine | up to 15 days
Rate and extent of excretion mass balance based on the total radioactivity in urine and faeces | up to 15 days
Cblood cells/Cplasma ratio of [14C]-radioactivity | up to 12 hours after drug administration
Cblood /Cplasma ratio of [14C]-radioactivity | up to 144 hours after drug administration
Identification of major metabolites in plasma, urine, and faeces | up to day 15
Cmax (maximum concentration of the analyte(s) in plasma) | up to 144 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte(s) in plasma) | up to 144 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte(s) in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 144 hours after drug administration
AUC0-inf. (area under the concentration-time curve of the analyte(s) in plasma over the time interval from 0 to infinity) | up to 144 hours after drug administration
λz (terminal rate constant in plasma) | up to 144 hours after drug administration
t1/2 (terminal half-life of the analyte(s) in plasma) | up to 144 hours after drug administration
MRTpo (mean residence time of the analyte(s) in the body after oral administration) | up to 144 hours after drug administration
CL/F (total clearance of the analyte in plasma after oral administration) | up to 144 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an oral dose) | up to 144 hours after drug administration
Ae0-tz (amount of analyte that is eliminated in urine within the time interval zero to tz, additionally excretion within each sampling interval will be calculated) | up to 15 days
fe0-tz (fraction of analyte excreted in urine within the time interval zero to tz in % of dose, additionally excretion within each sampling interval will be calculated) | up to 15 days
Aefaeces,0-tz (amount of analyte excreted in faeces within the time interval zero to tz, additionally excretion within each sampling interval will be calculated) | up to 15 days
fefaeces,0-tz (fraction of analyte excreted in faeces within the time interval zero to tz in % of dose, additionally excretion within each sampling interval will be calculated) | up to 15 days
CLR,t1-t2 (renal clearance of analyte from the within the time interval t1 to t2) | up to 15 days

SECONDARY OUTCOMES:
Number of patients with clinically relevant findings in vital signs | up to 23 days
Number of patients with clinically relevant findings in 12-lead electrocardiogram (ECG) | up to 23 days
Number of patients with clinically relevant laboratory findings | up to 23 days
Number of patients with adverse events | up to up to 44 days
Assessment of global tolerability on a 4-point scale | day 15